CLINICAL TRIAL: NCT02993445
Title: A Pilot Study on the Effect of Alternate Nostril Breathing and Foot Reflexology on Intraocular Pressure in Ocular Hypertension
Brief Title: Effect of Alternate Therapies on Intraocular Pressure in Ocular Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Temple University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 22105
Record Dates: First submitted 2016-12-08; First posted 2016-12-15 (Estimated); Results first posted 2020-11-27 (Actual); Last update posted 2020-11-27 (Actual); Status verified 2020-11

CONDITIONS: Ocular Hypertension
MeSH Terms: conditions — Ocular Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Alternate Nostril Breathing (Experimental): The procedure for ANB begins by bringing the right hand up to the nose; with the ring finger over the left nostril and the thumb over the right nostril, so that the nostrils may be closed by the fingers. The first step in the cycle is to hold the right nostril closed with the thumb, and exhale completely through the left nostril in a slow and controlled fashion, free from exertion and jerkiness. At the end of the exhalation, the patient will inhale slowly and completely back through the left nostril. At this point the patient will close the left nostril with the ring finger, open the right nostril by releasing the thumb, and repeat the exhale-inhale process through the right nostril, completing one cycle. Then the patient will switch back to the left nostril and begin the cycle again. This cycle will be performed for one session lasting approximately 5 minutes.
  Interventions: Other: Alternate Nostril Breathing
- Foot Reflexology (Experimental): The procedure for FR focuses on activating specific reflex areas on the foot linked with the eye and eye disease, via massage. Although in the interest of repeatable precision, we have decided to use a FR board (fig.1) to conduct the procedure. This board has two foot shaped pieces of wood mounted on a flat board with springs. On top of these wooden feet are small wooden nodes, which are organized at precise locations to activate the reflexology of the foot by stimulation certain pressure points. The patient will be instructed to rest their feet on these boards with a comfortable pressure for a period of 5 minutes.
  Interventions: Device: Foot Reflexology

INTERVENTIONS:
Other: Alternate Nostril Breathing
  Arms: Alternate Nostril Breathing
Device: Foot Reflexology
  Arms: Foot Reflexology

SUMMARY:
The purpose of this study is to evaluate the effect of complementary and alternative therapies, specifically alternate nostril breathing and foot reflexology, on intraocular pressure in patients with ocular hypertension.

DETAILED DESCRIPTION:
11 patients were recruited from Temple Ophthalmology between 2014 and 2016. Patients had ocular hypertension and were between the ages of 48-74. Patients were excluded if they currently performed ANB or FR, were unable to perform the task, had previous eye surgery or laser, were receiving other CAM for ocular hypertension, or were unable to complete a washout period. After a 30-day drug washout, patients completed either ANB or FR. After instruction, the assigned task was performed for 5 minutes. FR was done on a commercially available foot reflexology board (JAPAN TSUBO HH-700) focused at the base of the second and third toes of both feet. Two weeks later, patients completed the alternate task. IOP was measured before the task, immediately after the task and then every 30 minutes for two hours. Sign rank tests were used to evaluate IOP changes within and between each group.

ELIGIBILITY:
Inclusion Criteria:

* patients with ocular hypertension

Exclusion Criteria:

* currently performed alternate nostril breathing or foot reflexology
* were unable to perform the task
* had previous eye surgery or laser,
* were receiving other CAM for ocular hypertension
* were unable to complete a washout period if they using glaucoma eye drops

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2014-09; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Henderer, M.D., Principal Investigator — Temple University

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After a 30-day drug washout, patients were randomly assigned to complete either ANB or FR for 5 min. After instruction, patients completed either ANB or FR, and completed the alternate task 2 weeks later.
Units Other Than Participants: eyes
Groups:
- Alternate Nostril Breathing First, Then Foot Reflexology: The procedure for ANB begins by bringing the right hand up to the nose; with the ring finger over the left nostril and the thumb over the right nostril, so that the nostrils may be closed by the fingers. The first step in the cycle is to hold the right nostril closed with the thumb, and exhale completely through the left nostril in a slow and controlled fashion, free from exertion and jerkiness. At the end of the exhalation, the patient will inhale slowly and completely back through the left nostril. At this point the patient will close the left nostril with the ring finger, open the right nostril by releasing the thumb, and repeat the exhale-inhale process through the right nostril, completing one cycle. Then the patient will switch back to the left nostril and begin the cycle again. This cycle will be performed for one session lasting approximately 5 minutes.
  Patients will complete 2 week wash out and then return for foot reflexology.
  The procedure for FR focuses on activating specific reflex areas on the foot linked with the eye and eye disease, via massage. Although in the interest of repeatable precision, we have decided to use a FR board (fig.1) to conduct the procedure. The patient will be instructed to rest their feet on these boards with a comfortable pressure for a period of 5 minutes.
- Foot Reflexology First, Then Alternate Nostril Breathing: The procedure for FR focuses on activating specific reflex areas on the foot linked with the eye and eye disease, via massage. Although in the interest of repeatable precision, we have decided to use a FR board (fig.1) to conduct the procedure. The patient will be instructed to rest their feet on these boards with a comfortable pressure for a period of 5 minutes.
  Patients will complete 2 week wash out and then return for alternate nostril breathing.
  The procedure for ANB begins by bringing the right hand up to the nose; with the ring finger over the left nostril and the thumb over the right nostril, so that the nostrils may be closed by the fingers. The first step in the cycle is to hold the right nostril closed with the thumb, and exhale completely through the left nostril in a slow and controlled fashion, free from exertion and jerkiness. At the end of the exhalation, the patient will inhale slowly and completely back through the left nostril. At this point the patient will close the left nostril with the ring finger, open the right nostril by releasing the thumb, and repeat the exhale-inhale process through the right nostril, completing one cycle. Then the patient will switch back to the left nostril and begin the cycle again. This cycle will be performed for one session lasting approximately 5 minutes.
Period: First Intervention (5 Minutes)
Arm/Group | Alternate Nostril Breathing First, Then Foot Reflexology | Foot Reflexology First, Then Alternate Nostril Breathing
Started | 6; 12 eyes | 5; 10 eyes
Completed | 6; 12 eyes | 5; 10 eyes
Not Completed | 0; 0 eyes | 0; 0 eyes
Period: Washout (2 Weeks)
Arm/Group | Alternate Nostril Breathing First, Then Foot Reflexology | Foot Reflexology First, Then Alternate Nostril Breathing
Started | 6; 12 eyes | 5; 10 eyes
Completed | 6; 12 eyes | 5; 10 eyes
Not Completed | 0; 0 eyes | 0; 0 eyes
Period: Second Intervention (5 Mins)
Arm/Group | Alternate Nostril Breathing First, Then Foot Reflexology | Foot Reflexology First, Then Alternate Nostril Breathing
Started | 6; 12 eyes | 5; 10 eyes
Completed | 6; 12 eyes | 5; 10 eyes
Not Completed | 0; 0 eyes | 0; 0 eyes

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Alternate Nostril Breathing First, Then Foot Reflexology | Foot Reflexology First, Then Alternate Nostril Breathing | Total
Number analyzed (Participants) | 6 | 5 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.0 (9.69) | 65.4 (7.44) | 62.64 (8.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 3 | 2 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 3 | 6
  White | 3 | 2 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Corneal Thickness [Mean (Standard Deviation); unit: mm]
  Right Eye | 567.8 (36.78) | 572.7 (37.0) | 569.6 (34.21)
  Left Eye | 568.2 (39.7) | 575.3 (53.1) | 570.88 (41.49)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Intraocular Pressure (mmHg)
Description: Measurement of intraocular pressure after each treatment for 30min intervals for total of 2hours. Time points used in the calculation include baseline, 30 mins, 60 mins, 90 mins, and 120 mins.
Time Frame: 2 hours
Measure: Mean (Standard Deviation); unit: mm Hg
Units Other Than Participants: eyes
Groups:
- Alternate Nostril Breathing Alternate Nostril Breathing First, Then Foot Reflexology: The procedure for ANB begins by bringing the right hand up to the nose; with the ring finger over the left nostril and the thumb over the right nostril, so that the nostrils may be closed by the fingers. The first step in the cycle is to hold the right nostril closed with the thumb, and exhale completely through the left nostril in a slow and controlled fashion, free from exertion and jerkiness. At the end of the exhalation, the patient will inhale slowly and completely back through the left nostril. At this point the patient will close the left nostril with the ring finger, open the right nostril by releasing the thumb, and repeat the exhale-inhale process through the right nostril, completing one cycle. Then the patient will switch back to the left nostril and begin the cycle again. This cycle will be performed for one session lasting approximately 5 minutes.
  Patients will complete 2 week wash out and then return for foot reflexology. The procedure for FR focuses on activating specific reflex areas on the foot linked with the eye and eye disease, via massage. Although in the interest of repeatable precision, we have decided to use a FR board (fig.1) to conduct the procedure. The patient will be instructed to rest their feet on these boards with a comfortable pressure for a period of 5 minutes.
Arm/Group | Alternate Nostril Breathing Alternate Nostril Breathing First, Then Foot Reflexology | Foot Reflexology First, Then Alternate Nostril Breathing
Number analyzed (Participants) | 6 | 5
Number analyzed (eyes) | 12 | 10
mm Hg
  Baseline | 25.3 (1.61) | 26.8 (4.39)
  30 minutes IOP | 23.9 (2.19) | 22.5 (4.12)
  60 minutes IOP | 23.5 (2.35) | 22.7 (4.03)
  90 minutes IOP | 21 (2.66) | 22.5 (3.64)
  120 minutes IOP | 22.6 (2.9) | 25.3 (1.28)

2. Primary Outcome: Change From Baseline in Intraocular Pressure (mmHg)
Description: Measurement of intraocular pressure after each treatment for 30min intervals for total of 2hours. Time points used in the calculation include baseline, 30 mins, 60 mins, 90 mins, and 120 mins.
  This is after the 2 week washout period. Participants have switched interventions
Time Frame: 2 hours
Measure: Mean (Standard Deviation); unit: mm Hg
Units Other Than Participants: eyes
Arm/Group | Alternate Nostril Breathing Alternate Nostril Breathing First, Then Foot Reflexology | Foot Reflexology First, Then Alternate Nostril Breathing
Number analyzed (Participants) | 6 | 5
Number analyzed (eyes) | 12 | 10
mm Hg
  Baseline | 24.3 (2.22) | 26.5 (4.43)
  30 minutes IOP | 21.3 (2.00) | 23.9 (3.99)
  60 minutes IOP | 20.6 (2.00) | 23.45 (4.02)
  90 minutes IOP | 20.4 (2.08) | 22.7 (4.33)
  120 minutes IOP | 20.6 (2.23) | 22.7 (3.65)

ADVERSE EVENTS:
Time Frame: 1 hour after each task patients were assessed for adverse events
Groups:
- Alternate Nostril Breathing: The procedure for ANB begins by bringing the right hand up to the nose; with the ring finger over the left nostril and the thumb over the right nostril, so that the nostrils may be closed by the fingers. The first step in the cycle is to hold the right nostril closed with the thumb, and exhale completely through the left nostril in a slow and controlled fashion, free from exertion and jerkiness. At the end of the exhalation, the patient will inhale slowly and completely back through the left nostril. At this point the patient will close the left nostril with the ring finger, open the right nostril by releasing the thumb, and repeat the exhale-inhale process through the right nostril, completing one cycle. Then the patient will switch back to the left nostril and begin the cycle again. This cycle will be performed for one session lasting approximately 5 minutes.
  Alternate Nostril Breathing
- Foot Reflexology: The procedure for FR focuses on activating specific reflex areas on the foot linked with the eye and eye disease, via massage. Although in the interest of repeatable precision, we have decided to use a FR board (fig.1) to conduct the procedure. This board has two foot shaped pieces of wood mounted on a flat board with springs. On top of these wooden feet are small wooden nodes, which are organized at precise locations to activate the reflexology of the foot by stimulation certain pressure points. The patient will be instructed to rest their feet on these boards with a comfortable pressure for a period of 5 minutes.
  Foot Reflexology
Arm/Group | Alternate Nostril Breathing | Foot Reflexology
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 0/11 | 0/11

LIMITATIONS AND CAVEATS:
Small sample size; No control group

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes